CLINICAL TRIAL: NCT05708131
Title: Outcomes of Functional Substrate Mapping of Ventricular Tachycardia (Func-VT) - an International Propensity-matched Prospective Registry
Brief Title: Outcomes of Functional Substrate Mapping of Ventricular Tachycardia
Acronym: VTFM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: 315453
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this registry database is to demonstrate the safety and effectiveness of functional ventricular tachycardia (VT) ablation using SENSE protocol in patients with ischaemic VT. Mortality and the need for ICD therapies at 12 months post-ablation will be compared with propensity-matched controls undergoing substrate-based ablation alone.

DETAILED DESCRIPTION:
This is an international multicentre prospective registry. Participating centres will collect data during the pre-assessment, procedure, and follow-up visits at 6 and 12 months, according to standard practice. It is anticipated that the enrolment duration will be approximately 12 months, with the data being matched with that collected from a control group of patients undergoing conventional Ventricular tachycardia ablation methods.

ELIGIBILITY:
Inclusion Criteria:

One of the following VT events (within the last 6 months) + Ejection Fraction <40%:

A: ≥3 episodes of VT treated with anti-tachycardia pacing (ATP), at least one of which is symptomatic.

B: ≥1 appropriate ICD shock. C: ≥3 VT episodes within 24 hr. D: Sustained VT below the detection rate of the ICD.

Exclusion Criteria:

* Contraindication to VT ablation
* Renal failure (CrCl < 15 mL/min)
* NYHA IV or CCS IV angina
* STEMI within 1 month
* CABG within 3 months
* PCI within 1 month
* Pregnant
* Life expectancy < 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Composite of cardiovascular mortality and ICD therapy | 12 months
  Composite of cardiovascular mortality and implantable cardioverter-defibrillator (ICD) therapy

SECONDARY OUTCOMES:
Length of hospital stay | 1 month
  Length of hospital stay
Left ventricular function on echocardiogram | 6 months
  Left ventricular function on echocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Neil Srinvasan, MBBS, Principal Investigator — Mid and South Essex NHS FT
Locations (8):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States
- Onassis Cardiac Surgery Center, Athens, Greece
- Spain (2):
  - Virgen de las Nieves University Hospital, Granada
  - Arrhythmia Unit, University Hospital Ramón y Cajal, Madrid
- United Kingdom (4):
  - Basildon University Hospital, Basildon
  - Royal Sussex County Hospital, Brighton
  - Royal Brompton & Harefield hospital, London
  - St Bartholomew's Hospital, London